CLINICAL TRIAL: NCT00113698
Title: Trial of ACE Inhibition in Children With Mitral Regurgitation After Repair of AVSD
Brief Title: Angiotensin Converting Enzyme Inhibition in Children With Mitral Regurgitation
Acronym: AceiMR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lower than expected enrollment
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pediatric Heart Network (Other)
Responsible Party: Principal Investigator, Lois LuAnn Minich, Primary Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 185; U01HL068269 (NIH); U01HL068270 (NIH); U01HL068279 (NIH); U01HL068281 (NIH); U01HL068285 (NIH); U01HL068288 (NIH); U01HL068290 (NIH); U01HL068292 (NIH)
Record Dates: First submitted 2005-06-09; First posted 2005-06-10 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Heart Defects, Congenital; Heart Septal Defects, Ventricular; Heart Failure, Congestive
MeSH Terms: conditions — Heart Defects, Congenital; Heart Septal Defects, Ventricular; Heart Failure | interventions — Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Other: Placebo
- 2 (Active Comparator): Ace inhibition (enalapril)
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Enalapril — Up-titration period is to reach the highest tolerated dose up to a maximum of 0.4 mg/kg/day
  Arms: 2
Other: Placebo — Placebo An inert preparation with similar appearance and taste to the drug
  Arms: 1

SUMMARY:
This study will evaluate the efficacy and safety of angiotensin converting enzyme inhibition (ACE-I) therapy for the treatment of mitral regurgitation (MR).

DETAILED DESCRIPTION:
BACKGROUND:

MR causes volume overload and hemodynamic burden on the left ventricle. Initial compensatory mechanisms may fail, leading to increased severity. Patients who have had repair of an atrioventricular septal defect (AVSD) are selected for this study as they have a relatively high incidence of moderate MR and their regurgitant orifice is mobile and dynamic, contributing to the likelihood that they might respond to medical therapy.

DESIGN NARRATIVE:

This is a randomized, double-blind, placebo-controlled trial of ACE-I therapy in children less than 18 years of age with at least moderate MR who are at least 6 months postoperative from repair of an AVSD. A non-randomized Observational Phase enrolled 181 children who were less than 6 months postoperative from repair of an AVSD, who were then evaluated at 6 months for trial eligibility.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 18 years of age and at least 6 months post AVSD repair or reoperation
* At least moderate MR
* Asymptomatic or minimally symptomatic, defined by Ross Heart Failure Class I or II
* Atrioventricular synchrony (paced or intrinsic)

Exclusion Criteria:

* Tetrology of Fallot, total or partial anomalous venous connection
* More than trivial MS or outflow obstruction
* Other sources of LV volume overload
* Hypertrophic obstructive cardiomyopathy
* Significant residual coarctation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2004-12; Primary Completion 2005-11 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the effect of ACE-I therapy with that of placebo on left ventricular size | Measured after six months of therapy

SECONDARY OUTCOMES:
Comparison of the effect of ACE-I therapy with placebo on MR severity, left ventricular geometry, hemodynamics, and signs and symptoms of congestive heart failure | 6 months on study drug
Evaluation of the early natural history of MR in the six months after repair of an AVSD | 6 months on study drug
Comparison of the incidence of adverse events occurring in subjects treated with ACE-I therapy to that in subjects receiving placebo (measured after six months of therapy) | 6 months on safety drug

CONTACTS AND LOCATIONS:
Overall Officials: LuAnn Minich, MD, Principal Investigator — Primary Children's Hospital, Salt Lake City, UT
Locations (7):
- United States (6):
  - Children's Hospital Boston, Boston, Massachusetts
  - Columbia College of Physicians and Surgeons, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Primary Children's Hospital, Salt Lake City, Utah
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Li JS, Colan SD, Sleeper LA, Newburger JW, Pemberton VL, Atz AM, Cohen MS, Golding F, Klein GL, Lacro RV, Radojewski E, Richmond ME, Minich LL. Lessons learned from a pediatric clinical trial: the Pediatric Heart Network angiotensin-converting enzyme inhibition in mitral regurgitation study. Am Heart J. 2011 Feb;161(2):233-40. doi: 10.1016/j.ahj.2010.10.030. PMID 21315203
- [Derived] Atz AM, Hawkins JA, Lu M, Cohen MS, Colan SD, Jaggers J, Lacro RV, McCrindle BW, Margossian R, Mosca RS, Sleeper LA, Minich LL; Pediatric Heart Network Investigators. Surgical management of complete atrioventricular septal defect: associations with surgical technique, age, and trisomy 21. J Thorac Cardiovasc Surg. 2011 Jun;141(6):1371-9. doi: 10.1016/j.jtcvs.2010.08.093. Epub 2010 Dec 15. PMID 21163497